CLINICAL TRIAL: NCT03682302
Title: A Multicenter Study to Evaluate the Pharmacokinetics and Safety of EXPAREL for Postsurgical Analgesia in Pediatric Subjects Aged 6 to Less Than 17 Years
Brief Title: Multicenter Study for Pediatric Subjects Evaluating Pharmacokinetics and Safety of EXPAREL
Acronym: PLAY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-319
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Pain Management
Keywords: Pediatric
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: 12 to less than 17 years, undergoing spine surgery, EXPAREL (Experimental): Single dose of EXPAREL 4 mg/kg (not to exceed a maximum total dose of 266 mg) via local infiltration at the end of spine surgery.
  Interventions: Drug: Exparel
- Group 1: 12 to less than 17 years, undergoing spine surgery, bupivacine (Active Comparator): Single dose of bupivacaine hydrochloride (HCl) 2 mg/kg (not to exceed a maximum total dose of 175 mg) via local infiltration at the end of spine surgery.
  Interventions: Drug: 0.5% Bupivacaine HCl
- Group 2: 6 to less than 12 years, undergoing spine surgery, EXPAREL (Experimental): Single dose of EXPAREL 4 mg/kg (not to exceed a maximum total dose of 266 mg) via local infiltration at the end of spine surgery.
  Interventions: Drug: Exparel
- Group 2: 6 to less than 12 years, undergoing cardiac surgery, EXPAREL (Experimental): Single dose of EXPAREL 4 mg/kg (not to exceed a maximum total dose of 266 mg) via local infiltration at the end of cardiac surgery.
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Exparel — EXPAREL 4mg/kg (maximum 266 mg)
  Other Names: Liposomal bupivacaine
  Arms: Group 1: 12 to less than 17 years, undergoing spine surgery, EXPAREL; Group 2: 6 to less than 12 years, undergoing cardiac surgery, EXPAREL; Group 2: 6 to less than 12 years, undergoing spine surgery, EXPAREL
Drug: 0.5% Bupivacaine HCl — Bupivacaine HCl 2mg/kg
  Other Names: Bupivacaine
  Arms: Group 1: 12 to less than 17 years, undergoing spine surgery, bupivacine

SUMMARY:
Primary Objective: To evaluate the pharmacokinetics (PK) of EXPAREL in pediatric subjects aged 6 to less than 17 years undergoing various types of surgeries.

Secondary Objective: To evaluate the safety of EXPAREL in pediatric subjects aged 6 to less than 17 years undergoing various types of surgeries.

DETAILED DESCRIPTION:
This is a Phase 3, two-part, multi-center, open-label study designed to evaluate the PK and safety profile of EXPAREL in pediatric subjects aged 6 to less than 17 years when administered intraoperatively at the end of surgery via local infiltration. 90 pediatric subjects undergoing spine and/or cardiac surgeries are planned for enrollment.

Part 1 is a multicenter, randomized, open-label study in subjects aged 6 to less than 17 years undergoing spine or cardiac surgeries. There will be 2 treatment groups: Group 1 will include subjects aged 12 to less than 17 years, while Group 2 will include subjects aged 6 to less than 12 years

Part 2 is a multicenter, randomized, open-label, safety study in subjects aged 6 to less than 17 years undergoing spine or cardiac surgeries. There will be 2 treatment groups: Group 1 will include subjects aged 12 to less than 17 years, while Group 2 will include subjects aged 6 to less than 12 years.

Subjects will be screened within 30 days prior to study drug administration. During the screening visit, subjects will be assessed for past or present neurologic, cardiac, and general medical conditions that, in the opinion of the investigator, would preclude them from study participation.

Subjects will undergo their pre-planned spinal or cardiac surgeries per the institution's standard of care. On Day 1, eligible subjects will receive the study drug intraoperatively at the end of surgery via local infiltration into the surgical site. Dosing of EXPAREL will be based on body weight, with a starting dose of 4 mg/kg (maximum 266 mg).

There is no required length of stay in the hospital; subjects may be discharged based on the medical judgment of the treating physician.

A follow-up phone call will be scheduled for all subjects on Day 7. A final follow-up visit will be made on Day 30 to all subjects who would have received the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects whose parent(s) or guardian(s) has/have signed and dated the ICF for the subject to participate in the study, and subjects who have provided written assent to participate in the study (if capable).
2. American Society of Anesthesiologists (ASA) Class 1-3.
3. Male or female subjects 6 to less than 17 years of age on the day of surgery.
4. Body mass index (BMI) at screening within the 5th to 95th percentile for age and sex (see Appendix 5).
5. A negative pregnancy test for female subjects of childbearing potential must be available prior to the start of surgery. The pregnancy test must be conducted in the preoperative holding area according to the study site's standard of care.
6. Subjects and their parent(s)/guardian(s) must be able to speak, read, and understand the language of the ICF and any instruments used for collecting subject-reported outcomes to enable accurate and appropriate responses to study assessments, and provide informed consent/assent.
7. Subjects must be able to adhere to the study visit schedule and complete all study assessments.

Exclusion Criteria:

1. Currently pregnant, breastfeeding, or planning to become pregnant during the study or within 1 month after study drug administration.
2. History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics or to opioid medication.
3. Contraindication to bupivacaine HCl or other amide-type local anesthetics or to opioid medication.
4. Administration of EXPAREL or bupivacaine HCl within 30 days prior to study drug administration.
5. Subjects with coagulopathies or immunodeficiency disorders.
6. History of, suspected, or known addiction to or abuse of drugs or alcohol within the past 2 years.
7. Clinically significant medical or psychiatric disease that, in the opinion of the investigator, indicates an increased vulnerability to study drugs and/or procedures.
8. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

   In addition, the subject will be ineligible to receive study drug if he or she meets the following criterion during surgery:
9. Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postsurgical course.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igor Grachev, MD, PhD, Study Director — Pacira Pharmaceuticals, Inc
Locations (17):
- United States (17):
  - Loma Linda University, Loma Linda, California
  - Shriners Hospitals for Children, Northern California, Sacramento, California
  - Stanford University, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours / Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Nicklaus Children's Hospital, Miami, Florida
  - Shriners Hospitals for Children-Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - McGovern Medical School at UTHealth, Houston, Texas
  - Southwest Scoliosis Institute, Plano, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Tirotta CF, de Armendi AJ, Horn ND, Hammer GB, Szczodry M, Matuszczak M, Wang NQ, Scranton R, Ballock RT. A multicenter study to evaluate the pharmacokinetics and safety of liposomal bupivacaine for postsurgical analgesia in pediatric patients aged 6 to less than 17 years (PLAY). J Clin Anesth. 2021 Dec;75:110503. doi: 10.1016/j.jclinane.2021.110503. Epub 2021 Sep 14. PMID 34534923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 02 April 2019 and 24 September 2019 at 15 sites in the US (both Groups).
Groups:
- Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacine: Single dose of bupivacaine HCl 2 mg/kg (not to exceed a maximum total dose of 175 mg) via local infiltration at the end of spine surgery.
Period: Overall Study
Arm/Group | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, EXPAREL | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacine | Group 2: 6 to Less Than 12 Years, Undergoing Spine Surgery, EXPAREL | Group 2: 6 to Less Than 12 Years, Undergoing Cardiac Surgery, EXPAREL
Started | 31 | 30 | 6 (1 subject enrolled in Group 2, not treated, and surgery type unknown. Subject is not counted here.) | 30 (1 subject enrolled in Group 2, not treated, and surgery type unknown. Subject is not counted here.)
Completed | 30 | 28 | 5 | 28
Not Completed | 1 | 2 | 1 | 2
Not completed — Lost to Follow-up | 1 | 2 | 0 | 1
Not completed — Study drug was not administered | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population The Safety population consisted of all subjects who underwent the planned surgery and received study treatment, with analysis by actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, EXPAREL | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacine | Group 2: 6 to Less Than 12 Years, Undergoing Spine Surgery, EXPAREL | Group 2: 6 to Less Than 12 Years, Undergoing Cardiac Surgery, EXPAREL | Total
Number analyzed (Participants) | 31 | 30 | 5 | 29 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (1.33) | 13.9 (1.33) | 10 (1.73) | 8.7 (1.77) | 12.1 (2.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 2 | 14 | 66
  Male | 3 | 8 | 3 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 0 | 9 | 26
  Not Hispanic or Latino | 19 | 23 | 5 | 20 | 67
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 5 | 3 | 1 | 2 | 11
  White | 21 | 26 | 4 | 26 | 77
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 5 | 29 | 95
American Society of Anesthesiologists classification [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) classification was determined by physicians using the ASA Physical Status Classification System which assesses the patient's pre-anesthesia medical co-morbidities. ASA 1 patients would be considered a normal, healthy patient. ASA 2 is a patient with mild systemic disease (eg, smoker, well controlled diabetes or high blood pressure (HBP)). ASA 3 is a patient with severe systemic disease (eg poorly controlled diabetes or HBP). ASA 4 is a patient with severe systemic disease that is a constant threat to life (eg, recent myocardial infarction, stroke).
  Participants
    ASA 1 | 14 | 13 | 1 | 0 | 28
    ASA 2 | 16 | 13 | 2 | 2 | 33
    ASA 3 | 1 | 4 | 2 | 27 | 34

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-versus-time Curve (AUC) 0 to Infinity
Time Frame: 15, 30, 45 min, 1-1.25h, 2-4h, 10-18h, 24-36h, 42-60h (spine surgery) or 15, 30, 45 min, 1-1.25, 15-25, 20-40, 45-55, 64-72h (cardiac surgery)
Population: The pharmacokinetic population consisted of subjects who received study drug and provided at least 1 quantifiable plasma concentration, with analysis by actual treatment received.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, EXPAREL | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacine | Group 2: 6 to Less Than 12 Years, Undergoing Spine Surgery, EXPAREL | Group 2: 6 to Less Than 12 Years, Undergoing Cardiac Surgery, EXPAREL
Number analyzed (Participants) | 16 | 15 | 2 | 21
ng*h/mL | 14246.1 (9118.83) | 5709.4 (3281.74) | 11569.5 (7306.07) | 26164.0 (28038.35)

2. Primary Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, EXPAREL | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacine | Group 2: 6 to Less Than 12 Years, Undergoing Spine Surgery, EXPAREL | Group 2: 6 to Less Than 12 Years, Undergoing Cardiac Surgery, EXPAREL
Number analyzed (Participants) | 16 | 15 | 2 | 21
ng/mL | 357.3 (125.31) | 563.6 (320.93) | 319.5 (164.76) | 447.1 (243.41)

3. Primary Outcome: The Apparent Terminal Elimination Half-life (t1/2el)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, EXPAREL | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacine | Group 2: 6 to Less Than 12 Years, Undergoing Spine Surgery, EXPAREL | Group 2: 6 to Less Than 12 Years, Undergoing Cardiac Surgery, EXPAREL
Number analyzed (Participants) | 16 | 15 | 2 | 21
hours | 26.8 (21.26) | 8.4 (6.26) | 13.4 (4.60) | 24.9 (20.58)

4. Primary Outcome: Apparent Clearance (CL/F)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, EXPAREL | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacine | Group 2: 6 to Less Than 12 Years, Undergoing Spine Surgery, EXPAREL | Group 2: 6 to Less Than 12 Years, Undergoing Cardiac Surgery, EXPAREL
Number analyzed (Participants) | 16 | 15 | 2 | 21
Liters/hour | 17.5 (7.47) | 20.5 (8.27) | 14.5 (2.70) | 7.4 (3.20)

5. Primary Outcome: Apparent Volume of Distribution (Vd/F)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, EXPAREL | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacine | Group 2: 6 to Less Than 12 Years, Undergoing Spine Surgery, EXPAREL | Group 2: 6 to Less Than 12 Years, Undergoing Cardiac Surgery, EXPAREL
Number analyzed (Participants) | 16 | 15 | 2 | 21
Liters | 546.4 (269.42) | 226.8 (110.63) | 271.1 (43.58) | 216.1 (83.77)

6. Primary Outcome: Area Under the Plasma Concentration-versus-time Curve (AUC) 0 to Tlast
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, EXPAREL | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacine | Group 2: 6 to Less Than 12 Years, Undergoing Spine Surgery, EXPAREL | Group 2: 6 to Less Than 12 Years, Undergoing Cardiac Surgery, EXPAREL
Number analyzed (Participants) | 16 | 15 | 2 | 21
ng*h/mL | 9042.5 (3762.82) | 5232.9 (2538.37) | 10249.6 (5956.56) | 16776.4 (7935.80)

ADVERSE EVENTS:
Time Frame: Screening through postsurgical Day 14
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (eg, abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug without any judgment about causality.
  Serious AEs were defined as per clinicaltrials.gov.
Groups:
- Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacaine: Single dose of bupivacaine HCl 2 mg/kg (not to exceed a maximum total dose of 175 mg) via local infiltration at the end of spine surgery.
Arm/Group | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, EXPAREL | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacaine | Group 2: 6 to Less Than 12 Years, Undergoing Spine Surgery, EXPAREL | Group 2: 6 to Less Than 12 Years, Undergoing Cardiac Surgery, EXPAREL
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/5 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/5 | 2/29
Other Adverse Events (participants affected / at risk) | 19/31 | 22/30 | 5/5 | 9/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, EXPAREL (N=31) | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacaine (N=30) | Group 2: 6 to Less Than 12 Years, Undergoing Spine Surgery, EXPAREL (N=5) | Group 2: 6 to Less Than 12 Years, Undergoing Cardiac Surgery, EXPAREL (N=29)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Wound infection fungal (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, EXPAREL (N=31) | Group 1: 12 to Less Than 17 Years, Undergoing Spine Surgery, Bupivacaine (N=30) | Group 2: 6 to Less Than 12 Years, Undergoing Spine Surgery, EXPAREL (N=5) | Group 2: 6 to Less Than 12 Years, Undergoing Cardiac Surgery, EXPAREL (N=29)
Constipation (Gastrointestinal disorders) | 8 | 9 | 1 | 4
Nausea (Gastrointestinal disorders) | 10 | 6 | 1 | 2
Vomiting (Gastrointestinal disorders) | 9 | 5 | 1 | 4
Hypoesthesia oral (Gastrointestinal disorders) | 1 | 3 | 3 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 | 8 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Vision blurred (Eye disorders) | 4 | 3 | 3 | 1
Visual impairment (Eye disorders) | 2 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0
Hypoesthesia (Nervous system disorders) | 0 | 2 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 2 | 7 | 2 | 0
Anemia postoperative (Injury, poisoning and procedural complications) | 4 | 0 | 1 | 0
Delayed recovery from anesthesia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 4 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0
Hypoacusis (Ear and labyrinth disorders) | 2 | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results conducted at Site shall not be published before 1st multicenter publication by Sponsor but can proceed if there is no such publication ≤18 months after study completion/termination at all sites and all data have been received. Before submitting manuscript/materials to an outside person/entity, site shall give Sponsor 60 days to review and comment. Site shall, upon request, further delay publication/presentation for ≤120 days to allow Sponsor to protect its interests in Inventions.

DOCUMENTS (2):
  • Study Protocol (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03682302/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT03682302/SAP_001.pdf